CLINICAL TRIAL: NCT01534650
Title: Movement Disorder Quantification Algorithm Development
Status: Completed | Type: Observational
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GLNT-001
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Parkinson's Disease; Essential Tremor
Keywords: motion sensors; tremor; bradykinesia; gait; balance; dyskinesia
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Tremor; Hypokinesia; Dyskinesias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to collect kinematic motion data from subjects with movement disorders such as Parkinson's disease (PD) and essential tremor (ET) to develop and validate algorithms for quantifying motor symptoms such as tremor, bradykinesia (slowed movements), dyskinesias (sudden, involuntary movements), gait, and balance during standardized tasks and/or activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Clinical diagnosis of idiopathic Parkinson's disease or essential tremor
* Able to provide informed consent

Exclusion Criteria:

* Significant medical or psychiatric illness
* Not capable of following the required clinical instructions
* Serious medical conditions that compromise safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of Northeastern Ohio with a movement disorder such as Parkinson's disease or essential tremor.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2012-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Processed kinematics | During assessment
  Motion data collected during various motor tasks will be processed and compared to video review.

CONTACTS AND LOCATIONS:
Overall Officials: Dustin A Heldman, PhD, Principal Investigator — Great Lakes NeuroTechnologies Inc.
Locations (1):
- Great Lakes NeuroTechnologies Inc. Movement Disorders Laboratory, Valley View, Ohio, United States